CLINICAL TRIAL: NCT03668470
Title: Dulaglutide and Insulin MicrosecretiON in Type 1 Diabetes : A Randomized Double-blind Placebo-controlled Trial
Brief Title: Dulaglutide and Insulin MicrosecretiON in Type 1 Diabetes
Acronym: DIAMOND GLP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL18_0047
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Adult Subjects With Type1Diabetes and Insulin Microsecretion
Keywords: type 1 diabetes; insulin microsecretion; dulaglutide; randomized; double-blind placebo-controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: Multicentric, investigator-initiated, randomized, double-blinded, therapeutic clinical trial, placebo-controlled, two arm parallel group intervention trial during 24 weeks, phase II.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dulaglutide (Experimental): Experimental group receiving 1.5 mg Dulaglutide subcutaneously weekly in addition to their usual insulin regimen during 24 weeks
  Interventions: Drug: Dulaglutide
- placebo (Placebo Comparator): Control group receiving placebo subcutaneously weekly in addition to their usual insulin regimen during 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Dulaglutide 1.5mg : One injection per week during 24 weeks
  Arms: Dulaglutide
Drug: Placebo — Placebo: one injection per week during 24 weeks
  Arms: placebo

SUMMARY:
Some patients with type 1 diabetes (T1D) can still have some remaining insulin-positive cells in the pancreas and secrete little amounts of insulin. Despite the presence of residual beta cells, the HbA1C levels remain at high levels due to functional defects of insulin secretion associated with glucotoxicity. Previous trials have indicated that treatment with a Glucagon-like peptide 1 (GLP-1 )receptor agonist in T1D with some residual beta-cell function might improve glycemic control, reduce dose of insulin and risk of hypoglycemia.

The general hypothesis of DIAMOND-GLP1 is that GLP1-R agonists will improve blood glucose

After initial screening to select insulin microsecretors and a run-in period of one month, patients will be randomized into two arms and followed in parallel for 24 weeks :

* Experimental group receiving 1.5 mg Dulaglutide s.c weekly in addition to their usual insulin regimen
* Control group receiving placebo s.c weekly in addition to their usual insulin regimen.

The primary endpoint is HbA1c value at 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with T1D> 4years, with age range 20-60years
* Diabetes onset after the age of 15years
* Duration of diabetes <15 years
* Treated with continuous sub-cutaneous insulin infusions (CSI) or multiple daily injections of insulin (MDI)
* Measuring their blood sugar at least four times daily
* Glycated hemoglobin (HbA1C) at screening >7 and <10%
* 16.0 kg/m2 <BMI<30.0kg/m2
* Patients with childbearing potential should use effective contraception, defined as methods with a failure rate ≤ 2 % per year (OMS 2011) during the study.
* Patients who gave its written informed consent to participate to the study
* Patients affiliated to a social insurance regime

Randomization criteria:

Patients with fasting ultra-sensitive (us) C-peptide above 15pmol/l

Exclusion Criteria:

* Patients are not eligible for this study if any of the following exclusion criteria apply:
* Patients with type 2 diabetes (T2D)
* Hypersensitivity to dulaglutide and/or any of its excipients
* Subjects with history of severe hypoglycemia or recent (< 6 months) history of diabetic ketoacidosis
* History of gastrointestinal disease with prolonged (> 3 months) nausea or vomiting, liver or kidney diseases, pancreatitis, thyroid medullary cancer or familial history of multiple endocrine neoplasia type 2
* Estimated glomerular filtration rate<60ml/min/ 1.73m2 (CKD-EPI method)
* Congestive heart failure
* Any uncontrolled disease, cancers essentially
* Chronic use of paracetamol containing products, which may falsely raise sensor glucose readings
* Use of tricyclic antidepressant, selective serotonin reuptake inhibitor, triptans, neuroleptic drugs and glucocorticoid.
* Patient who participated in another clinical trial on experimental drug in the previous 30 days
* Patients of childbearing potential who are not using adequate contraception; Female patients who are pregnant or lactating.
* Gastric bypass surgery
* Patients under guardianship

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
HbA1c level | after 24 weeks of treatment
  Blood level

SECONDARY OUTCOMES:
AUC us C-peptide following a MMT | before and after 24 weeks of treatment
  Evaluation and comparison before and after 24wks of treatment with Dulaglutide vs placebo the area under curve (AUC) of ultrasensitive (us) C-peptide response from 6 values following a mixed meal test (MMT)
Glucagon levels fasting and following a MMT | before and after 24 weeks of treatment
  Evaluation and comparison before and after 24wks of treatment with Dulaglutide vs placebo AUC glucagon from 6 values on fasting and after MMT
AUC us C-peptide over AUC blood glucose levels following a MMT | before and after 24 weeks of treatment
  Evaluation and comparison the ratio of the area under curve (AUC) of us C-peptide over the glucose response following a mixed meal test (MMT) with before and after 24 weeks of treatment Dulaglutide vs placebo
Daily percent times spent with continuous glucose measurements (CGM) readings between 4 and 10mmol/l, above and below this range | the run-in period (1 month) and after 24 weeks of treatment
  Evaluation and comparison the changes in the daily percent time spent with continuous glucose measurements (CGM) readings between 4 and 10mmol/l during the run-in period (1 month) and after 24 weeks with Dulaglutide vs placebo, coefficients of variation (CV) and standard deviation values (SD) as well as the average daily risk change (ADRR) of glucose values to assess blood glucose variability.
Daily insulin doses and basal/ prandial ratio | : before and after 24weeks of treatment
  Evaluation and comparison before and after 24wks of treatment with Dulaglutide vs placebo the daily insulin doses and basal/ prandial ratio
: Body weight | before and after 24weeks of treatment
% carbohydrates | the run-in period (1 month) and after 24 weeks of treatment
  Evaluate and compare the changes in mean carbohydrate intake during the run-in period and after 24 weeks with Dulaglutide vs placebo
Number of symptomatic hypoglycemic episodes | 20 months
  Evaluation and comparison the number of symptomatic (both minor and severe) hypoglycemic episodes with Dulaglutide vs placebo during the study
Number of adverse events | 20 months
  Evaluation and comparison the number of adverse events with Dulaglutide vs placebo during the study
Autoantibodies to GAD65 | : before and after 24wks of treatment
  Evaluation and comparison before and after 24wks of treatment the levels and subtypes of autoantibodies associated with T1D with and without dulaglutide
insulin doses : basal/ prandial ratio | before and after 24weeks of treatment
  the insulin basal/ prandial ratio
Autoantibodies to IA-2 | before and after 24wks of treatment
  Evaluation and comparison before and after 24wks of treatment the levels and subtypes of autoantibodies associated with T1D with and without dulaglutide
Autoantibodies to ZnT8 | before and after 24wks of treatment
  Evaluation and comparison before and after 24wks of treatment the levels and subtypes of autoantibodies associated with T1D with and without dulaglutide
coefficients of variation (CV) | the run-in period (1 month) and after 24 weeks of treatment
  coefficients of variation (CV) of daily percent times spent with continuous glucose measurements (CGM) readings between 4 and 10mmol/l, above and below this range .

CONTACTS AND LOCATIONS:
Overall Officials: Charles THIVOLET, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Service d'Endocrinologie, Maladies Métaboliques et Nutrition, CHU Grenoble, Hopital de la Tronche, La Tronche
  - Département d''Endocrinologie, Diabétologie, Nutrition ; CHU Montpellier ; Hôpital Lapeyronie, Avenue du Doyen Giraud, Montpellier
  - Service d'Endocrinologie, Maladies Métaboliques et Nutrition,CHU Nantes,Hôpital Nord Laennec,Bd Jacques-Monod,Saint-Herblain, Nantes
  - Service de Diabétologie et Maladies Métaboliques, Assistance Publique des Hôpitaux de Paris ;Hôpital Cochin, 27 rue du Faubourg Saint-Jacques, Paris
  - Service d'Endocrinologie, Diabétologie, Maladies de la Nutrition, Hospices Civils de Lyon, Centre hospitalier Lyon-Sud, Pierre-Bénite
  - Service de Diabétologie Maladies Métaboliques et Nutrition ; CHU Toulouse, Pôle cardiovasculaire et métabolique, Hôpital Rangueil ; 1, avenue du Professeur Jean Poulhès - TSA 50032, Toulouse
  - Service de Diabétologie, Maladies Métaboliques, Nutrition ; CHU Nancy ; Technopôle Nancy-Brabois ; Rue du Morvan,, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided